CLINICAL TRIAL: NCT01853631
Title: Phase I Study of Activated T-Cells Expressing Second or Third Generation CD19-Specific Chimeric Antigen Receptors for Advanced B-Cell Non-Hodgkin's Lymphoma, Acute Lymphocytic Leukemia and Chronic Lymphocytic Leukemia (SAGAN)
Brief Title: Activated T-Cells Expressing 2nd or 3rd Generation CD19-Specific CAR, Advanced B-Cell NHL, ALL, and CLL (SAGAN)
Acronym: SAGAN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-31970 SAGAN; SAGAN (Other: Baylor College of Medicine)
Record Dates: First submitted 2013-05-01; First posted 2013-05-15 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Acute Lymphocytic Leukemia
Keywords: chronic Lymphocytic Leukemia; refractory; recurrent; aggressive B-cell Lymphoma; CD19; Non-Hodgkin Lymphoma; CD28; CD137; 4-1BB; acute lymphocytic leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation: CD19 CAR T Cells for B-cell ALL (Experimental): Each patient will receive a dose of CD19 CAR T Cells administered as an infusion. Each infusion will consist of CD19.CAR/28 T cells and CD19.CAR/28137 T cells.
  Interventions: Genetic: Dose Escalation Phase:CD19.CAR/28 and CD19.CAR/28137 T cells
- Dose Expansion: CD19 CAR T Cells for B-cell ALL (Experimental): Each patient will receive the maximum tolerated dose (MTD) of CD19 CAR T Cells administered as an infusion. Each infusion will consist of CD19.CAR/28 T cells and CD19.CAR/28137 T cells.
  Interventions: Genetic: Expansion Phase: CD19.CAR/28 and CD19.CAR/28137 T cells
- Dose Escalation: CD19 CAR T Cells for B-cell NHL/CLL (Experimental): Each patient will receive a dose of CD19 CAR T Cells administered as an infusion. Each infusion will consist of CD19.CAR/28 T cells and CD19.CAR/28137 T cells.
  Interventions: Genetic: Dose Escalation Phase:CD19.CAR/28 and CD19.CAR/28137 T cells
- Dose Expansion: CD19 CAR T Cells for B-cell NHL/CLL (Experimental): Each patient will receive the maximum tolerated dose (MTD) of CD19 CAR T Cells administered as an infusion. Each infusion will consist of CD19.CAR/28 T cells and CD19.CAR/28137 T cells.
  Interventions: Genetic: Expansion Phase: CD19.CAR/28 and CD19.CAR/28137 T cells

INTERVENTIONS:
Genetic: Dose Escalation Phase:CD19.CAR/28 and CD19.CAR/28137 T cells — Three dose levels will be evaluated.
  Group 1: CD19.CAR/28137ζ at 1×10^6 cells/m^2 and CD19.CAR/28ζ at 1×10^6 cells/m^2
  Group 2: CD19.CAR/28137ζ at 5×10^6 cells/m^2 and CD19.CAR/28ζ at 5×10^6 cells/m^2
  Group 3: CD19.CAR/28137ζ at 2×10^7 cells/m^2 and CD19.CAR/28ζ at 2×10^7 cells/m^2
  Arms: Dose Escalation: CD19 CAR T Cells for B-cell ALL; Dose Escalation: CD19 CAR T Cells for B-cell NHL/CLL
Genetic: Expansion Phase: CD19.CAR/28 and CD19.CAR/28137 T cells — The primary goal of the expanded cohort is to further study the safety profiles of CAR-T cells in each of the disease settings, both with or without lymphodepleting chemotherapy given before CAR-T cell infusion.
  Arms: Dose Expansion: CD19 CAR T Cells for B-cell ALL; Dose Expansion: CD19 CAR T Cells for B-cell NHL/CLL

SUMMARY:
Subjects on this study have a type of lymph gland cancer called Non-Hodgkin Lymphoma, acute lymphocytic leukemia, or chronic Lymphocytic Leukemia (these diseases will be referred to as "lymphoma" or "leukemia"). The lymphoma or leukemia has come back or has not gone away after treatment.

The body has different ways of fighting infection and disease. No one way seems perfect for fighting cancers. This research study combines two different ways of fighting disease, antibodies and T cells, hoping that they will work together. Both antibodies and T cells have been used to treat patients with cancer. They have shown promise, but have not been strong enough to cure most patients.

T cells can kill tumor cells but normally there are not enough of them to kill all the tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person.

The antibody used in this study is called anti-CD19. It first came from mice that have developed immunity to human lymphoma. This antibody sticks to lymphoma cells because of a substance on the outside of these cells called CD19. CD19 antibodies have been used to treat people with lymphoma and leukemia. For this study, anti-CD19 has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor.

In the laboratory, the investigators found that T cells work better if they also add proteins that stimulate T cells, such as one called CD28. Adding the CD28 makes the cells last longer in the body but not long enough for them to be able to kill the lymphoma cells. The investigators believe that if they add an extra stimulating protein, called CD137, the cells will have a better chance of killing the lymphoma cells.

The investigators are going to see if this is true by putting the CD19 chimeric receptor with CD28 alone into half of the cells and the CD19 chimeric receptor with CD28 and CD137 into the other half of the cells. These CD19 chimeric receptor T cells with CD28 and with or without CD137 are investigational products not approved by the FDA.

The purpose of this study is to find the biggest dose of chimeric T cells that is safe, to see how long the T cell with each sort of chimeric receptor lasts, to learn what the side effects are and to see whether this therapy might help people with lymphoma or leukemia.

DETAILED DESCRIPTION:
Patients will give the investigators blood to make CD19 CD28 (with and without CD137) chimeric receptor-T cells in the laboratory. These cells will be grown and frozen. To make the T cells, investigators will take blood (or blood from a donor) and stimulate it with growth factors to make the T cells grow. To get the CD19 antibody and CD28 (with or without CD137) to attach to the surface of the T cell, they will insert the antibody gene into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps to find the T cells in the blood after injecting them; in order to tell them apart investigators have made two viruses that are slightly different because one has CD137. These two viruses can be told apart by a special laboratory test. Because the patient will receive cells with a new gene in them, the patient will be followed for a total of 15 years to see if there are any long term side effects of gene transfer. If the patient cannot visit the clinic, he or she will be contacted by the research coordinator or physician.

When subjects enroll on this study, they will be assigned a dose of CD19 chimeric receptor-T cells. Several studies suggest that the infused T cells need room to be able to proliferate and accomplish their functions and that this may not happen if there are too many other T cells in circulation.

Because of that, if the subject's level of circulating T cells is relatively high, s/he may receive one treatment of cyclophosphamide (Cytoxan) and fludarabine if the doctor thinks this is appropriate. This drug will decrease the numbers of the subject's own T cells before infusion of the CD19 chimeric receptor T cells. If subject is already receiving chemotherapy, this may not be needed. The investigators would prefer subjects do not receive other chemotherapy until 6 weeks after cell infusion but they can do so if their doctor thinks it is medically necessary.

Patients will be given an injection of cells into the vein through an IV at the assigned dose. The injection will take about 20 minutes. The investigators will follow them in the clinic after the injection for up to 3 hours.

If after a 6 week evaluation period after the infusion, the patient seems to be experiencing a benefit (confirmed by radiological studies, physical exam and/or symptoms), s/he may be able to receive up to five additional doses of the T cells if s/he wishes. The first repeat infusion can only take place at least 6 weeks after the first infusion. Any additional infusions after that would be at least 4 weeks apart. All additional infusions will be at the same dose level received the first time or a lower dose. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

ELIGIBILITY:
Inclusion Criteria:

PROCUREMENT

Referred patients (or respective donors) will initially be consented for procurement of blood for generation of the transduced ATL. Eligibility criteria at this stage include:

* Diagnosis of recurrent B-cell lymphoma or leukemia (ALL or CLL), or newly diagnosed patients unable to receive or complete standard therapy OR diagnosis of relapsed/refractory aggressive B-cell lymphoma with a treatment plan that will include high dose therapy and autologous stem cell transplantation.
* CD19-positive tumor (result can be pending at this time).
* Age <= 75 years. The first 3 patients treated on the study should be adults (>= 18 years).
* Hgb greater than or equal to 7.0 (can be a transfused value)
* If pheresis required to collect blood:
* Creatinine < 1.5 x upper limit normal
* AST <1.5 × upper limit normal
* PT and APTT <1.5 × upper limit normal
* Informed consent explained to, understood by and signed by patient/guardian (and donor, where applicable). Patient/guardian given copy of informed consent.

TREATMENT

* Diagnosis of recurrent B-cell lymphoma leukemia (ALL or CLL), or newly diagnosed patients unable to receive or complete standard therapy OR diagnosis of relapsed/refractory aggressive B-cell lymphoma with a treatment plan that will include high dose therapy and autologous stem cell transplantation.
* CD19-positive tumor.
* Age <= 75 years. The first 3 patients treated on the study should be adults (>= 18 years).
* Bilirubin less than 3 times the upper limit of normal.
* AST less than 5 times the upper limit of normal.
* Estimated GFR > 50 mL/min
* Pulse oximetry of > 90% on room air
* Karnofsky or Lansky score of > 60%.
* Recovered from acute toxic effects of prior chemotherapy at least one week before entering this study. PD1/PDL1 inhibitors will be allowed if medically indicated.
* Available autologous or syngeneic activated peripheral blood T cell products (CD28ζ and CD28/CD137ζ) with more than or equal to 15% expression of CD19.CAR determined by flow cytometry.
* Life expectancy of greater than 12 weeks.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
* Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.

Exclusion Criteria:

PROCUREMENT

* Active infection requiring antibiotics.
* No history of other cancer (except non-melanoma skin cancer or in situ breast cancer or cervix cancer) unless the tumor was successfully treated with curative intent at least 2 years before trial entry.

TREATMENT

* Currently receiving any investigational agents or received any tumor vaccines within the previous 6 weeks. (Note treatment with PD1/PDL1 inhibitors is allowed.)
* History of hypersensitivity reactions to murine protein-containing products.
* Pregnant or lactating.
* Tumor in a location where enlargement could cause airway obstruction.
* Active infection with HIV or HTLV.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-02; Primary Completion 2026-12 (Estimated); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity (DLT) | 6 weeks
  Toxicity will be evaluated according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) scale, version 4. DLT will be defined as any of the following that is NOT (1) pre-existing, or (2) due to infection (to which patients with CLL and NHL are predisposed), or (3) due to underlying malignancy, and that may, after consultation with the FDA when indicated, be considered possibly, probably, or definitely related to the study cellular products: (1) Non-hematologic DLT is any grade 3 or grade 4 non-hematologic toxicity, including allergic reactions to T cell infusions; (2) Hematologic DLT is defined as any grade 4 hematologic toxicity. Patients with evidence of bone marrow disease (metastases or diffuse infiltration) are not evaluable for hematologic dose limiting toxicity.

SECONDARY OUTCOMES:
Survival of CD19.CAR-ATLs | 15 years
  Survival will be measured by a real time Q-PCR assay to detect CD19.CAR-ATLs in peripheral blood from subjects. Plots will be generated to depict patterns of survival. Also, longitudinal modeling techniques will be used.
Frequency of the two distinct T cell products post infusion | 15 years
  To compare the changes in frequency of two different T-cell products in the same patient, two different Q-PCR assays will be used, which distinguish each CAR by the presence or absence of the CD137 co-stimulatory endodomain gene.
Number of patients with tumor response | 15 years
  Tumor responses will be assessed by the International Working Group Revised Response Criteria for Malignant Lymphoma or the National Cancer Institute CLL Working Group Recommendations, as applicable.
Percentage of circulating modified T cells after additional doses | 15 years
  Changes in the percentage of circulating modified T cells after additional doses will be measured by each respective real time Q-PCR assay to detect CD19.CAR-ATLs in peripheral blood from subjects. Plots will be generated to depict patterns of survival. Also, longitudinal modeling techniques will be used.
Function of CD19.CAR-ATLs | up to 15 years
  To study the function of CD19.CAR-ATLs, the following assays will be performed on PBMCs isolated from subjects: (1) ELISPOT for interferon-gamma release using CD19-positive cells and CD19-negative target cells; (2) Other functional assays, such as in vitro reactivation of PBMCs, in patients on whom the appropriate reagents are available; and (3) Immunophenotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo M, Zhang H, Zhu L, Xu Q, Gao Q. CAR-T Cell Therapy: Challenges and Optimization. Crit Rev Immunol. 2021;41(1):77-87. doi: 10.1615/CritRevImmunol.2021037253. PMID 33822526